CLINICAL TRIAL: NCT05411237
Title: A Phase III, Randomized, Open-Label, Non-Inferiority Study of Paclitaxel and Pegylated Liposomal Doxorubicin for Treatment of HIV-related Kaposi Sarcoma in Resource-Limited Settings
Brief Title: Paclitaxel and Pegylated Liposomal Doxorubicin for Treatment of HIV-related Kaposi Sarcoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC-114; U01CA121947 (NIH)
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Kaposi Sarcoma; HIV-1-infection; AIDS-related Kaposi Sarcoma
Keywords: Paclitaxel; Pegylated liposomal doxorubicin; AIDS associated Kaposi Sarcoma; Human Immunodeficiency Virus; HIV-related Kaposi Sarcoma
MeSH Terms: conditions — Sarcoma, Kaposi; AIDS-related Kaposi sarcoma; Acquired Immunodeficiency Syndrome | interventions — liposomal doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pegylated Liposomal Doxorubicin (Active Comparator): Participants will receive a single intravenous dose of PLD 20 mg/m2 once every 3 weeks for a total of 18 weeks.
  Interventions: Drug: Pegylated liposomal doxorubicin
- Paclitaxel (Active Comparator): Participants will receive a single intravenous dose of PTX 100 mg/m2 once every 3 weeks for a total of 18 weeks.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — PLD 20 mg/m2 on Day 1 of every 21-day cycle
  Other Names: Doxil
  Arms: Pegylated Liposomal Doxorubicin
Drug: Paclitaxel — PTX 100 mg/m2 on Day 1 of every 21-day cycle
  Other Names: Taxol
  Arms: Paclitaxel

SUMMARY:
This study is being done to determine if two different anti-cancer drugs, paclitaxel (PTX) and pegylated liposomal doxorubicin (PLD) have similar effects on treating Kaposi Sarcoma (KS) in people living with HIV (human immunodeficiency virus) in sub-Saharan Africa. Patients with HIV-related KS will receive either PTX or PLD once every 3 weeks for a total of six cycles.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection.
2. Histologically confirmed KS at any time prior to study entry, confirmed by an AIDS Malignancy Consortium (AMC)-certified pathologist.
3. Current stage T1 KS (irrespective of prior treatment with antiretroviral therapy (ART) OR

   Stage T0 KS that has progressed or not responded after a minimum of 12 weeks of treatment with ART. Participants with T0 KS must have either:
   * 20 or more skin and/or oral KS lesions, and/or
   * any number of lesions on exposed body areas that have an adverse effect on quality of life (e.g., stigmatization).
4. Men and women ≥ 18 years. Because no dosing or adverse event data are currently available on the use of PTX or PLD for AIDS-KS in persons <18 years of age, children are excluded from this study
5. Karnofsky performance status ≥ 60 (ECOG ≤ 2).
6. Echocardiogram or Multiple gated acquisition scanning (MUGA) showing an ejection fraction ≥ 50%.
7. Ability and willingness of participant or legal guardian to provide informed consent.
8. Participants may be ART-naïve or ART-experienced but must be able to receive an ART regimen considered likely to result in HIV suppression.
9. Measurable cutaneous KS, defined as follows:

   * When available, a minimum of five bi-dimensionally measurable KS cutaneous marker lesions.
   * If fewer than five bi-dimensionally measurable marker lesions are available, the total surface area of the marker lesion(s) must be ≥ 700mm2.
10. The following laboratory values obtained within 14 days prior to study entry:

    * Absolute Neutrophil Count ≥ 1000 cells/mm3.
    * Hemoglobin ≥ 8 g/dL (may be achieved with transfusion if clinically indicated, in the opinion of the investigator).
    * Platelet count ≥ 75,000/mm3.
    * ALT, AST, Alkaline phosphatase < 5 × upper limit of normal (ULN).
    * Total bilirubin: ≤ 1.5 × ULN, unless the participant is receiving an antiretroviral drug known to be associated with increased bilirubin, in which case the direct fraction should be ≤ 2 x the ULN.
    * Creatinine < institutional ULN OR estimated glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
11. Women of reproductive potential, defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months), must have a negative pregnancy test done within 24 hours of initiating the protocol-specified chemotherapy medication.
12. Participants must agree to use two reliable forms of contraception simultaneously while receiving study protocol-specified medication and for 6 months after stopping the medication.
13. Adequate venous access.
14. No prior chemotherapy or use of systemic cytotoxic therapy agents.
15. Participant is able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

1. Current acute, chronic, or recurrent infections that are serious, in the opinion of the site investigator, for which the participant has not completed at least 14 days of therapy before study entry and/or is not clinically stable.
2. Serious illness necessitating hospitalization/systemic treatment within 14 days prior to study entry
3. Breastfeeding or pregnant women are excluded because of potential risks of cytotoxic chemotherapy to an unborn child or infant.
4. Known history of congestive heart failure and/or systolic ejection fraction < 50%.
5. Prior radiotherapy to KS indicator lesions
6. Prior or current immunotherapy
7. Any immunomodulator, HIV vaccine, live attenuated vaccine, other investigational vaccine within 30 days prior to study entry, excluding vaccines against COVID-19/SARS-CoV-2, which are permitted.
8. Known allergy/hypersensitivity to the study drug or its formulation
9. Any condition, including the presence of laboratory abnormalities, which in the opinion of the responsible investigator places the subject at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study.
10. Corticosteroid use at doses above those given for replacement therapy for adrenal insufficiency within the last 30 days prior to study entry.
11. Patients with psychiatric illness and/or social circumstances that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 48 weeks | 48 weeks
  Progression free survival (PFS) is defined as the length of time from enrollment into the study until disease progression or death. Disease progression will be assessed using the Kaposi Sarcoma Response Evaluation Criteria. Progressive disease is defined as: 1) 25% increase in the sum of perpendicular diameters of the indicator lesions; 2) 25% increase in the total number of KS lesions or the appearance of 5 new lesions; OR 3) 25% increase in the number of raised lesions

SECONDARY OUTCOMES:
Frequency and severity of adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 in participants receiving PLD or PTX. | 96 weeks
  The frequency of adverse events that occur in patients receiving PLD will be compared with the frequency of adverse events in patients receiving PTX
Objective response rate for AIDS-related KS in patients receiving PLD and PTX | 96 weeks
  The objective response rate is defined as the sum of the number of complete and partial responses in patients receiving PLD or PTX.
Duration of Response in patients receiving PLD and PTX | 96 weeks
  Response duration is defined as the time from first documentation of complete or partial response as measured by KS response criteria to the documentation of first progression of disease as measured by KS response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Susan Krown, MD, Study Chair — AIDS Malignancy Consortium

REFERENCES:
- [Derived] Chapola JC, Kleber SL, Krown SE, Painschab M. Cost-effectiveness protocol for treating adult HIV-infected patients with Kaposi sarcoma in resource-limited settings: a phase III, randomized, open-label, non-inferiority study of paclitaxel and pegylated liposomal doxorubicin. Cost Eff Resour Alloc. 2025 Nov 24;23(1):78. doi: 10.1186/s12962-025-00677-x. PMID 41286911